CLINICAL TRIAL: NCT01552837
Title: Effects of Quetiapine on Ultrastructural Hippocampal and Neurochemical Changes in Patients With Bipolar Disorder: Searching for Antidepressant and Mood Stabilising Neurophysiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1449L00030; 2007-000479-40 (EudraCT Number); EK 024/07 (Other: Ethics Commettee Number); 07-010 (Other: Sponsor's Code)
Record Dates: First submitted 2012-03-02; First posted 2012-03-13 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Bipolar Disorder
Keywords: Diffusion Tensor Imaging,; quetiapine; Bipolar Disorder; hippocampus; Volume Brain Morphometry; Magnetic Resonance Spectroscopy; effect of quetiapine on hippocampal neurogenesis
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy volunteers (No Intervention): MRI compatible, no present or past DSM-IV diagnosis
- patients with Bipolar Disorder (Active Comparator): MRI compatible, presence of DSM-IV diagnosis for Bipolar Disorder
  Interventions: Drug: Seroquel

INTERVENTIONS:
Drug: Seroquel — for 4 weeks, 300 - 800 mg per day in 2 doses
  Arms: patients with Bipolar Disorder

SUMMARY:
The aim of the study was to determine the pharmacological induced equivalents of neurogenesis and synaptic sprouting in the hippocampus, localized volume changes, changes in water content and neurochemical changes in the medial temporal regions.

DETAILED DESCRIPTION:
Quetiapine is an antipsychotic that has mood stabilizing and antidepressant effects (Vieta, 2005). Animal studies showed that the expression of neurotrophins and the subsequent modulation of the neuroplastic processes, including neurogenesis in the hippocampus, play a key role in the mechanism of mood stabilizing (Kim et al., 2004) and antidepressant (Santarelli et al., 2003). Since atypical antipsychotics also have antidepressant and mood stabilizing effect, it is hypothesized that the common mechanism of action in all three pharmacological classes is neurogenesis and synaptic sprouting in the hippocampal region. Thus, the aim of this study was to test this hypothesis.

Quetiapine was associated with antidepressant and mood stabilizing effects in patients with bipolar disorder (Vieta, 2005). The evidence based on animal studies shows that administration of quetiapine attenuates the decrease in levels of brain-derived neurotrophic factor in the hippocampi. This may explain the improved cognitive symptoms in patients with schizophrenia and depression (Luo et al., 2005, Park et al, 2006).

The aim of the study was to determine the pharmacological induced equivalents of neurogenesis and synaptic sprouting in the hippocampus, localized volume changes, changes in water content and neurochemical changes in the medial temporal regions.

ELIGIBILITY:
Inclusion Criteria:

* age ranging 18 - 55 years old
* intelligence coefficient (IQ) of minimum 85 as estimated by MWT-B
* MRI compatibility
* for healthy volunteers - no DSM-IV diagnosis
* patients should have had a diagnosis of bipolar disorder in accordance with DSM-IV.

Exclusion Criteria:

* substances or alcohol abuse or dependence (except caffeine and nicotine) at enrollment;
* medical conditions that would affect absorption, distribution, metabolism or excretion of study treatment;
* unstable or inadequately treated medical illness (diabetes, angina, pectoris, hypertension);
* diabetes mellitus
* patients who in the opinion of the investigator pose a risk of suicide or danger to self or others,
* patients who known intolerance or lack of response to Quetiapine fumarate,
* patients who use of any of the cytochrome P450 3A4 inhibitors (ketoconazole, itraconazole, nelfinavir, ritonavir, fluvoxamine and saquinavir) in the 14 days preceding enrollment,
* patients who use of any of the cytochrome P450 inducers (phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort and glucocorticoids) in the 14 days preceding enrollment,
* current treatment of Quetiapine or use of mood stabilizer or antidepressant as co-medication throughout the study.
* lack of inform consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2007-12; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Anisotropy in hippocampal formation detected with Diffusion Tensor Imaging (DTI) | after 6 weeks
  Detection of pharmacologically induced equivalents of neurogenesis and synaptic sprouting in the hippocampal region.

SECONDARY OUTCOMES:
safety and tolerability of medical treatment | every time during the study
  Observation of adverse events and tolerability assessed by vital signs and clinical chemistry
Detection of pharmacologically induced localised volume changes | after 6 weeks
  Measurement with 3D MPRAGE (structural scan)
Detection of pharmacologically induced localised changes in water content | after 6 weeks
  differentiation between neurogenesis/sprouting and mere water intake
Detection of pharmacologically induced neurochemical changes in the medial temporal regions (Glx and NAA, choline) | after 6 weeks
  Measurement of glutamate and N-acetylaspartate in the medial temporal lobe with MRS
Detection of pharmacologically induced differential activation during an episodic memory task measured with fMRI. | after 6 weeks
  Measurement of BOLD response using fMRI during an episodic memory test

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Mathiak, Prof MD, Study Director — Department of Psychiatry, Psychotherapy and Psychosomatics, University Hospital Aachen
Locations (1):
- Department of Psychiatry, Psychotherapy and Psychosomatics, University Hospital Aachen, Aachen, Germany

REFERENCES:
- [Background] Basser PJ, Mattiello J, LeBihan D. Estimation of the effective self-diffusion tensor from the NMR spin echo. J Magn Reson B. 1994 Mar;103(3):247-54. doi: 10.1006/jmrb.1994.1037. PMID 8019776
- [Background] Luo C, Xu H, Li XM. Quetiapine reverses the suppression of hippocampal neurogenesis caused by repeated restraint stress. Brain Res. 2005 Nov 23;1063(1):32-9. doi: 10.1016/j.brainres.2005.09.043. Epub 2005 Nov 4. PMID 16271709
- [Background] Vieta E. Mood stabilization in the treatment of bipolar disorder: focus on quetiapine. Hum Psychopharmacol. 2005 Jun;20(4):225-36. doi: 10.1002/hup.689. PMID 15880391